CLINICAL TRIAL: NCT00310661
Title: A Dual-centre, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Determine the Effects of Various Adjunctive Doses of Sarizotan in the Treatment of Patients With Neuroleptic-induced Tardive Dyskinesia
Brief Title: Sarizotan in the Treatment of Neuroleptic-induced Tardive Dyskinesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Gary Remington, MD, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 005/2004
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Neuroleptic-induced Tardive Dyskinesia
Keywords: sarizotan; neuroleptic-induced tardive dyskinesia
MeSH Terms: interventions — sarizotan; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo hard gelatin capsules matching the investigational medication
  Interventions: Other: Placebo
- Sarizotan HCI (Experimental): Sarizotan HCI is administered at various doses ranging from 2-7mg.
  Interventions: Drug: Sarizotan

INTERVENTIONS:
Drug: Sarizotan — The dose of sariztan HCI for each patient in the drug arm will be given 2mg b.i.d. orally during the first 4 weeks of treatment. If efficacy is inadequate and there are no safety concerns, the option to raise the dose to 5mg b.i.d is given. After 8 weeks of treatment, the option to raise the dose to 7mg bid is given. Dose may remain the same or may be decreased again to the previous dose.
  Other Names: Sarizotan HCI
  Arms: Sarizotan HCI
Other: Placebo — Placebo for each patient randomized to the placebo arm will be given placebo (oral, twice daily) in a pill form for 12 weeks
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
TD is a troublesome and potentially irreversible side effect associated with the use of neuroleptics. While the newer neuroleptics are improved in this regard, they all still carry the risk of TD.

The present study proposes that sarizotan is a potential agent for treating neuroleptic-induced TD based on preliminary data indicating efficacy in the management of dyskinesias associated with Parkinson's disease. Its efficacy is further substantiated by pre-clinical data obtained from the vacuous chewing movement (VCM) model in rats, a model we employ ourselves in investigating the relationship between D2 occupancy and TD. The present study also examines the effects of sarizotan on cognitive function, given the association between TD and cognitive deficits.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the safety and the anti-dyskinetic properties of sarizotan at various dosages for neuroleptic-induced TD.

The secondary objective of the study is to assess the effects of sarizotan on cognitive function in patients with neuroleptic-induced TD.

The diagnosis of neuroleptic-induced TD will be confirmed by history and physical examination. Patients will be evaluated at baseline, 2, 4, 8, and 12 weeks. Safety will be assessed by vital signs, ECG, routine blood tests, the ACTH stimulation test, and the clinician's and patient's global impression of tolerability.

Procedures:

For efficacy, the primary outcome variable will be changes in the Abnormal Involuntary Movement Scale (AIMS), and a baseline score of >3 ('moderate') will be required for item 8 (Severity of Abnormal Movements). Quantitative evaluation of movements will be carried out in two ways. The first involves a series of instrumental and clinical measures that were developed as a battery for the assessment of antipsychotic-induced parkinsonism and TD. The second means of quantifying the movements involves the use of video recording, with independent evaluation by several raters (Appendix I). Such approaches have gained popularity in the quantification of movement disorders as a means of improving reliability.

Secondary measures will include the positive and negative syndrome scale (PANSS) and other movement disorder scales (Simpson-Angus Rating Scales) for acute extrapyramidal symptoms (EPS), and the Barnes Akathisia Rating Scale (BARS). Global impressions of efficacy and tolerability by the clinician (CGI) and by the patients (PGI) will be recorded at all study visits after the commencement of treatment. To assess potential cognitive changes that may occur in conjunction with TD changes, a battery of neuropsychological tests will be carried out at baseline and endpoint (see Appendix II). To assess the relationship with primary negative symptoms such as the deficit syndrome, the total and sub-scales of the Positive and Negative Syndrome Scale will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets the Schooler and Kane Diagnostic Criteria (25) for Tardive Dyskinesia as established by history and physical examination.
* a score of 3 or above for item 8 of the AIMS scale (Severity of Abnormal Movements) at baseline.
* For female patients: either the patient is surgically sterile, has been post-menopausal for at least 12 months, or she is using a reliable method of contraception (single-barrier methods alone will not be considered sufficiently reliable) and provides a negative pregnancy test at the screening visit.
* on a stable dose of his/her current antipsychotic (either typical or atypical) and movement disorder medication (e.g. anticholinergics) for at least one month before randomisation. For depot antipsychotics, this period will be at least one dosing interval.
* The patient gives full written informed consent for participation in the study.
* The patient has a level of understanding of English or Tamil sufficient to communicate effectively with the investigator and study staff, and to be able to complete the computerised neurocognitive test battery where necessary

Exclusion Criteria:

* Exclusion criteria listed in the Research Criteria for Tardive Dyskinesia as defined in DSM-IV (symptoms not due to another neurological or general medical condition such as Huntington's disease, Sydenham's chorea, spontaneous dyskinesia, hyperthyroidism, Wilson's disease, ill-fitting dentures, exposure to other medications causing acute reversible dyskinesia such as L?dopa or bromocriptine).
* Evidence of pre-existing tic disorders, neuroleptic-induced acute dystonia or neuroleptic-induced acute akathisia
* Risk of suicide (in the opinion of the investigator).
* Any of the following non-permitted concomitant medication: Metoclopramide in the 4 weeks before screening, Buspirone in the 4 weeks before screening, Azole antifungals (particularly ketoconazole), Etomidate, HIV proteinase inhibitors (e.g. indinavir, ritonavir), any tricyclic antidepressant in the 4 weeks before screening (SSRI antidepressants if at a stable dosage are permitted), Fludrocortisone, Intermittent therapy with oral corticoids, continuous therapy with <7.5mg/day (oral) prednisolone or an equivalent dose of a different corticoid (patients on continuous long-term therapy with a dose of >7.5mg prednisolone or equivalent may participate but should not undergo an ACTH challenge test).
* Treatment with electroconvulsive therapy within six months before the first study visit.
* Known history of drug dependence (except nicotine and caffeine) or alcohol dependence within the six months before the study (three months for known drug abuse).
* Evidence of any clinically significant endocrine, cardiac, renal, neurological, cerebrovascular, metabolic, gastrointestinal, immunological, allergic or respiratory disease. Patients who are not euthyroid.
* asthma or known hypersensitivity to antipsychotic drugs or ACTH
* Pregnancy or lactation.
* Any abnormal laboratory test result(s) of potential clinical significance at screening, including: Aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) greater than 3 ´ upper limit of normal (ULN), Creatinine >2 ´ ULN, total bilirubin >2 ´ ULN
* Participation in another clinical study within the 30 days before the first visit of the present study.
* Plasma cortisol concentration below 18 µg/dL 60 minutes after stimulation with 250 µg ACTH1-24 (for procedure see Section 7.9). (NOTE: This exclusion criterion is waived, and the test should not be carried out, for patients on continuous long-term therapy with a dose of >7.5mg prednisolone or equivalent.
* Lack of legal capacity, or limited legal capacity.)
* Known previous diagnosis of learning disability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-12; Primary Completion 2006-09 (Actual); Study Completion 2008-03

PRIMARY OUTCOMES:
Degree of change in the Abnormal Involuntary Movement Scale | 12 weeks

SECONDARY OUTCOMES:
Change in PANSS | 12 weeks
Change in Simpson-Angus Rating Scales for acute EPS | 12 weeks
Change in Barnes Akathisia Rating Scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Remington, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada
- Schizophrenia Research Foundation of India, Chennai, India

REFERENCES:
- [Background] Kleven MS, Barret-Grevoz C, Bruins Slot L, Newman-Tancredi A. Novel antipsychotic agents with 5-HT(1A) agonist properties: role of 5-HT(1A) receptor activation in attenuation of catalepsy induction in rats. Neuropharmacology. 2005 Aug;49(2):135-43. doi: 10.1016/j.neuropharm.2005.02.005. Epub 2005 Apr 1. PMID 15996562
- See also: CAMH web site — http://camh.net